CLINICAL TRIAL: NCT04209673
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Alleviation in Perioperative Fracture Patients
Brief Title: TENS and Perioperative Fracture Patients
Acronym: TENS
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082259; 05-19-16E (Other: Atrium)
Record Dates: First submitted 2019-12-13; First posted 2019-12-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-06

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transcutaneous nerve stimulation (TENS) patients: Patients who received a TENS unit after surgery
  Interventions: Other: Multimodal Pain management including TENS unit
- No TENS: Historic controls- Patients who did not receive a TENS unit after surgery
  Interventions: Other: Multimodal Pain management not including TENS unit

INTERVENTIONS:
Other: Multimodal Pain management including TENS unit — Patient receiving multimodal pain management strategies which includes the use of TENS.
  Groups: Transcutaneous nerve stimulation (TENS) patients
Other: Multimodal Pain management not including TENS unit — Patient receiving multimodal pain management strategies which does not includes the use of TENS.
  Groups: No TENS

SUMMARY:
This is a pilot study designed to evaluate the effectiveness of TENS as part of post-operative pain management. Subjects receiving a TENS unit as part of clinical practice will be approached for consent and followed for 12 months.

DETAILED DESCRIPTION:
Transcutaneous electrical nerve stimulation (TENS) is an affordable and non-invasive option for post-operative analgesia. Broadly, TENS devices deliver pulsed electrical impulses across skin to modulate pain. They are theorized to work through different mechanisms at multiple physiologic levels. Centrally, TENS units activate small-diameter sensory afferents (Aδ nerve fibers), which in turn activate descending pain-inhibitory networks. Peripherally, TENS activation of both large- and small-diameter sensory afferents blocks nociceptive signals to the brain and is instead perceived as TENS-induced paresthesias. Finally, TENS efficacy may also be mediated by µ-opioid, 5-hydroxytryptamine (HT)-1, and 5-HT-2 receptors, particularly at low-frequency electrical activity.2

There are inconclusive results for the adjunctive use of TENS to modulate pain, largely because of a relative paucity of high-quality trials and significant inter-study heterogeneity due to non-standardized protocols. Moreover, most studies within the orthopaedic literature have been concentrated primarily within the total knee arthroplasty (TKA) literature and may have limited generalizability to orthopaedic trauma patients. Some studies have shown a trend towards decreased opioid consumption with the adjunctive use of TENS (vs. placebo-TENS or standard care)3,4 while other studies have shown no difference in pain scores in the post-operative period.5-8 To the investigator's knowledge, only two recent randomized clinical trial (RCT)s have been conducted on non-TKA orthopaedic populations, both of which show promise for the use of TENS postoperatively. One prospective double-blind randomized trial on arthroscopic rotator cuff repairs found a 25% reduction in post-operative opioid consumption when TENS was used adjunctively for pain control .9 Another single-blind prospective RCT on Colles' fractures reported greater postoperative pain improvements in patients receiving TENS vs. placebo.10

There is a growing body of evidence to suggest that TENS therapy can reduce post-operative pain after orthopedic procedures. More high-quality studies are needed to strengthen this suggestion and to characterize specific protocols, populations, and orthopedic conditions for which it might work best. Transcutaneous electrical nerve stimulation, if shown to be effective, stands to serve as an affordable non-opioid, non-invasive option for the safe and effective treatment of pain in the orthopaedic trauma patient population.

TENS units are a non-significant risk device and, therefore, do not require an investigational device exemption (IDE) based upon FDA guidance.15-17 The sensor pads will be placed at the same time as the surgical fixation of the study injury. It does not present a potential serious risk to the health and welfare of patients.

Specific Aim 1: To pilot the use of TENS among a postoperative lower extremity injury population as part of multimodal pain management.

Null Hypothesis (H0): TENS cannot be delivered safely among this population. Alternative Hypothesis (HA): TENS can be delivered safely among this population.

Specific Aim 2: To compare utilization of inpatient and outpatient pain medications of patients treated with TENS and historical controls.

H0: Patients treated with TENS will require the same amount of opioids as historical controls.

HA: Patients treated with TENS will require less opioids (lower morphine milligram equivalent - MME) than historical controls during hospitalization and throughout 3-month follow up.

Specific Aim 3: To compare patient-reported outcomes of patients treated with TENS and historical controls.

H0 1: Patients treated with TENS will experience equivalent patient-reported outcomes as compared to historical controls.

HA 1: Patients treated with TENS will experience greater improvement in patient-reported outcomes (PROMIS 29) relative to baseline as compared to historical controls.

H0 2: Patients treated with TENS will report higher pain scores as compared to historical controls.

HA 2: Patients treated with TENS will report equivalent or lower pain scores as compared to historical controls.

This will be a prospective observational study of patients undergoing operative treatment of lower extremity conditions, including fracture fixation, treatment of nonunion, and deformity correction. The study will be conducted at a single Level I trauma center. Enrolled patients will receive TENS postoperatively during hospitalization; TENS units will also be sent home with patients for use throughout recovery. This group will be compared to controls injury-matched from a prospectively collected, historical database on mobility who did not receive treatment with TENS.

ELIGIBILITY:
Inclusion Criteria:

* Operative treatment of lower extremity conditions, including fracture fixation, treatment of nonunion, and deformity correction
* Injury or deformity of the femur, tibia (plateau, shaft, pilon), or hindfoot and ankle
* Isolated injury
* Age 18 years or older
* Able to provide consent

Exclusion Criteria:

* • Unable to provide consent (no use of LAR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective observational study of patients undergoing operative treatment of lower extremity conditions, including fracture fixation, treatment of nonunion, and deformity correction. The study will be conducted at a single Level I trauma center. Enrolled patients will receive TENS postoperatively during hospitalization; TENS units will also be sent home with patients for use throughout recovery. This group will be compared to controls injury-matched from a prospectively collected, historical database on mobility who did not receive treatment with TENS.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Opioid use | 3 months following TENS unit placement
  Total amount of opioid use calculated by converting all opiates to Morphine Milligram Equivalents

SECONDARY OUTCOMES:
Change in patient-reported outcomes measurement information system (PROMIS 29) scores | baseline and 3 months
  The PROMIS-29 assesses seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to participate in social roles and activities. Each of the seven domains has four questions which are scored on a five-point Likert scale. The PROMIS-29 scales will be scored using a T-score metric method available at the Assessment Center website (http://assessmentcenter.net). A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores mean more of the specific scale's construct, which may indicate a desirable or an undesirable outcome.

OTHER OUTCOMES:
Process Measures and Feasibility as measured by patient compliance- Usage | 3 months
  Number of times the TENS unit was used each day by patients
Process Measures and Feasibility as measured by patient compliance- Duration | 3 months
  The duration of each TENS unit session as measured in minutes
Process Measures and Feasibility as measured by patient compliance-Frequency/amplitude | 3 months
  The average frequency/amplitude of electrical current for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Department of Orthopaedic Surgery, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Li J, Song Y. Transcutaneous electrical nerve stimulation for postoperative pain control after total knee arthroplasty: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2017 Sep;96(37):e8036. doi: 10.1097/MD.0000000000008036. PMID 28906393
- [Background] Tedesco D, Gori D, Desai KR, Asch S, Carroll IR, Curtin C, McDonald KM, Fantini MP, Hernandez-Boussard T. Drug-Free Interventions to Reduce Pain or Opioid Consumption After Total Knee Arthroplasty: A Systematic Review and Meta-analysis. JAMA Surg. 2017 Oct 18;152(10):e172872. doi: 10.1001/jamasurg.2017.2872. Epub 2017 Oct 18. PMID 28813550
- [Background] Beckwee D, Bautmans I, Swinnen E, Vermet Y, Lefeber N, Lievens P, Vaes P. A systematic review investigating the relationship between efficacy and stimulation parameters when using transcutaneous electrical nerve stimulation after knee arthroplasty. SAGE Open Med. 2014 Jun 16;2:2050312114539318. doi: 10.1177/2050312114539318. eCollection 2014. PMID 26770730
- [Background] Mahure SA, Rokito AS, Kwon YW. Transcutaneous electrical nerve stimulation for postoperative pain relief after arthroscopic rotator cuff repair: a prospective double-blinded randomized trial. J Shoulder Elbow Surg. 2017 Sep;26(9):1508-1513. doi: 10.1016/j.jse.2017.05.030. Epub 2017 Jul 20. PMID 28735847
- [Background] Lee CH, Lee TY, Her JS, Liao WL, Hsieh CL. Single-Blinded, Randomized Preliminary Study Evaluating the Effect of Transcutaneous Electrical Nerve Stimulation on Postoperative Pain in Patients with Colles' Fracture. J Altern Complement Med. 2015 Dec;21(12):754-8. doi: 10.1089/acm.2015.0119. Epub 2015 Oct 23. PMID 26496205
- [Background] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Background] Seymour RB, Leas D, Wally MK, Hsu JR; PRIMUM Group. Prescription reporting with immediate medication utilization mapping (PRIMUM): development of an alert to improve narcotic prescribing. BMC Med Inform Decis Mak. 2016 Aug 22;16(1):111. doi: 10.1186/s12911-016-0352-x. PMID 27549364
- [Background] Garland D, Holt P, Harrington JT, Caldwell J, Zizic T, Cholewczynski J. A 3-month, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of a highly optimized, capacitively coupled, pulsed electrical stimulator in patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2007 Jun;15(6):630-7. doi: 10.1016/j.joca.2007.01.004. Epub 2007 Feb 15. PMID 17303443
- [Background] Deyo RA, Walsh NE, Martin DC, Schoenfeld LS, Ramamurthy S. A controlled trial of transcutaneous electrical nerve stimulation (TENS) and exercise for chronic low back pain. N Engl J Med. 1990 Jun 7;322(23):1627-34. doi: 10.1056/NEJM199006073222303. PMID 2140432
- [Background] U. S. Food and Drug Administration/Center for Devices and Radiological Health. (2006). Information Sheet Guidance For IRBs, Clinical Investigators, and Sponsors Significant Risk and Nonsignificant Risk Medical Device Studies : FDA public health advisory. Silver Spring, MD.
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Rakel BA, Zimmerman BM, Geasland K, Embree J, Clark CR, Noiseux NO, Callaghan JJ, Herr K, Walsh D, Sluka KA. Transcutaneous electrical nerve stimulation for the control of pain during rehabilitation after total knee arthroplasty: A randomized, blinded, placebo-controlled trial. Pain. 2014 Dec;155(12):2599-2611. doi: 10.1016/j.pain.2014.09.025. Epub 2014 Sep 28. PMID 25270585
- [Result] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Result] Jones I, Johnson MI. Transcutaneous electrical nerve stimulation. Continuing Education in Anaesthesia Critical Care & Pain. 2009;9(4):130-135.